CLINICAL TRIAL: NCT05075122
Title: Phase 2 Multicenter Study Investigating the Tolerability and Efficacy of UV1 Vaccine in Patients With Recurrent or Metastatic PD-L1 Positive (CPS≥1) Head and Neck Squamous Cell Carcinoma Planned for First-line Treatment With Pembrolizumab
Brief Title: Tolerability and Efficacy of UV1 Vaccine in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma Planned for First-line Treatment With Pembrolizumab
Acronym: FOCUS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: Ultimovacs ASA (Industry); Apotheke der Universitätsmedizin der Johannes Gutenberg-Universität Mainz (Germany) (Unknown); Axel Hinke. CCRC Cancer Clinical Research Consulting (Düsseldorf, Germany (Unknown)
Responsible Party: Principal Investigator, Mascha Binder, MD, Prof. Dr. med., Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KKSH176; 2020-005910-17 (EudraCT Number)
Record Dates: First submitted 2021-07-21; First posted 2021-10-12 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — sargramostim; Injections; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccination arm (Experimental): Pembrolizumab flat dose iv every 3 weeks + UV1 vaccination (UV1 plus GM-CSF/Sargramostim as adjuvant per vaccination)
  Interventions: Biological: UV1; Drug: Sargramostim for Injection; Drug: Pembrolizumab injection
- Calibration arm (Other): Pembrolizumab flat dose iv every 3 weeks
  Interventions: Drug: Pembrolizumab injection

INTERVENTIONS:
Biological: UV1 — UV1 vaccination (300 μg) UV1 vaccination will be applied in a dense schedule with three vaccinations during one week before initiation of pembrolizumab, followed by 5 additional vaccinations every 3 weeks on d1 of each cycle (5 cycles in total, duration of treatment will be 13 weeks in total, regular EOT at week 14)
  Arms: Vaccination arm
Drug: Sargramostim for Injection — 75 μg GM-CSF as adjuvant per vaccination. Applied in a dense schedule with three injections during one week before initiation of pembrolizumab, followed by 5 additional injections every 3 weeks on d1 of each cycle (5 cycles in total, duration of treatment will be 13 weeks in total, regular EOT at week 14).
  Arms: Vaccination arm
Drug: Pembrolizumab injection — 200mg flat dose iv every 3 weeks. Pembrolizumab will be administered beyond the EOT visit at physician discretion until disease progression and up to a maximum of two years (standard of care)

SUMMARY:
The primary objective of this study is to determine the clinical performance of UV1 vaccination as add on to standard pembrolizumab treatment in patients with recurrent or metastatic PD-L1 positive (CPS >=1) head and neck squamous cell carcinoma. Secondary objectives are to determine the efficacy in terms of overall survival ,objective response rate and duration of response. Moreover, this study will explore patient subgroups most likely deriving benefit from a targeted immunotherapy approach combining a checkpoint inhibitor with a cancer vaccine and help to establish liquid biopsy tumor monitoring in HNSCC.

DETAILED DESCRIPTION:
Overall survival of patients with metastatic or recurrent HNSCC has improved over the past decade but remains poor overall. Median overall survival is limited to less than 15 months, with the current standard of care (immune checkpoint blockade with or without chemotherapy). Many patients with HNSCC are frail and therefore cannot tolerate chemotherapy, reducing their treatment options to checkpoint inhibitor. Therefore, the development of effective and tolerable combination regimens is urgently needed, especially in first-line therapy. The FOCUS study will evaluate such a combination regimen in patients with metastatic or recurrent HNSCC. The experimental regimen evaluated in this study will test the first-line standard drug pembrolizumab in combination with the novel UV1 cancer vaccine. In the comparator arm, patients receive pembrolizumab as the standard of care. The aim is to assess whether the addition of UVI can increase the efficacy of the checkpoint inhibitor. Based on currently available data, a decrease in efficacy due to the combination of standard first-line therapy with pembrolizumab is unlikely. The FOCUS study could therefore establish a new 1st-line regimen with increased efficacy and acceptable tolerability, which would need to be compared with the standard of care in a larger phase III trial. Based on the biomarker data from the FOCUS study, a subsequent Phase 3 study would potentially test the regimen only in subpopulations with increased response probability. From the perspective of the individual patient, participants may benefit from the experimental combination through improved efficacy. On the other hand, this is a novel combination study for HNSCC, and there is a risk that efficacy may not improve.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a non-resectable recurrent or metastatic head and neck squamous cell carcinoma (not necessarily reconfirmed at time of enrolment)
* At least one measurable tumor lesion as per RECIST v1.1, (Scan not older than 4 weeks before randomization)
* Eligible for pembrolizumab monotherapy (PD-L1 CPS >/= 1% and adequate laboratory parameters for pembrolizumab monotherapy as assessed by the investigator)
* ECOG-performance score 0-2
* Written informed consent obtained according to international guidelines and local laws
* Ability to understand and give informed consent.
* Safe contraception measures for males and females. Procedures with a pearl index of less than 1% apply as safe pregnancy prevention measures.

Exclusion Criteria:

* Patients for whom a combination therapy of a checkpoint inhibitor and a chemotherapy is deemed necessary in the opinion of the investigator
* Participation in another interventional study simultaneously and within the last 30 days prior to inclusion (registries or observational studies allowed)
* Concurrent malignancies other than disease under study within 5 years prior to inclusion, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) treated with expected curative outcome
* Active, known, or suspected autoimmune disease requiring systemic treatment.
* A concomitant therapy with systemic immune suppression: use of chronic systemic steroid medication (up to 5 mg/day prednisolone equivalent is allowed; patients using physiological replacement doses of prednisone for adrenal or pituitary insufficiency are eligible)
* History of severe autoimmune disorder or history of organ transplant
* Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the subject to receive study drug.
* Significant acute or chronic infections including, among others (test not older than 4 weeks prior to randomization): Any positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS), Any positive test result for hepatitis B virus or hepatitis C virus indicating acute or chronic infection.
* Pregnancy or lactation
* (Bacterial) infections requiring systemic antibiotic treatment within 2 weeks prior to first dose of study treatment (depending on group assignment: either prior to first UV1 or prior to first pembrolizumab administration).
* History of allergy or hypersensitivity to study drug or human granulocyte-macrophage colony stimulating factor, yeast-derived products or any constituent of the products
* Receipt of a live vaccine within 30 days prior to start of therapy
* Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities.
* Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical study and therefore cannot form a rational intention in the light of the facts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rate | 6 months after first administration of study medication
  according to iRECIST

SECONDARY OUTCOMES:
Progression free survival | every three months, until progression of disease, maximum 12 months from the date of LPI (last patient in)
  according to iRECIST
Overall survival | every three months, until death, maximum 12 months from the date of LPI (last patient in)
Objective Response Rate | every three months, until death, maximum 12 months from the date of LPI (last patient in)
  Complete Remission (CR) + Partial Remission (PR) according to iRECIST
Duration of Response | every three months, until death, maximum 12 months from the date of LPI (last patient in)
  according to iRECIST
Rate of immune responses against hTERT peptides | Baseline, up to 8 weeks, time of progression (max. 12 months after LPI)
  measured by 3H-Thymidine proliferation and IFNgamma ELISPOT assays
Rate of clearance of ctDNA from blood on treatment | Baseline, week 5, week 8 and 1, 3, 6 months after EOT (max. 14 weeks), time of progression (max. 12 months after LPI)
Adverse Events | 3 months after EOT (maximum 25 weeks after start of treatment)
  according to NCI CTC AE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Mascha Binder, MD, Principal Investigator — University Medical Center Halle, Department of Hematology and Oncology
Locations (10):
- Germany (10):
  - Universitätsklinikum Aachen, Klinik für Hämatologie, Onkologie, Hämostaseologie, Aachen
  - Charité Universitätsmedizin, Comprehensive Cancer Center, Medizinische Klinik m.S. Hämatologie, Onkologie und Tumorimmunologie, Berlin
  - Universitätsklinikum Greifswald, Klinik für Hals-, Nasen-, Ohrenkrankheiten, Kopf- und Halschirurgie, Greifswald
  - Universitätsklinikum Halle (Saale), Klinik und Poliklinik für Innere Medizin IV, Halle
  - Universitätsklinikum Hamburg, Universitäres Cancer Center Hamburg UCCH, Hubertus Wald Tumorzentrum, Hamburg
  - Klinikum St. Georg gGmbH, Leipzig
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für HNO Heilkunde, Leipzig
  - Universitätsklinikum Mainz, III. Medizinische Klinik und Poliklinik, Mainz
  - Klinikum Stuttgart, Klinik für Hämatologie, Onkologie und Palliativmedizin, Stuttgart
  - Universitätsklinikum Würzburg, Comprehensive Cancer Center Mainfranken, Würzburg

REFERENCES:
- [Derived] Paschold L, Schultheiss C, Schmidt-Barbo P, Klinghammer K, Hahn D, Tometten M, Schafhausen P, Blaurock M, Brandt A, Westgaard I, Kowoll S, Stein A, Hinke A, Binder M. Inflammation and limited adaptive immunity predict worse outcomes on immunotherapy in head and neck cancer. NPJ Precis Oncol. 2025 Aug 5;9(1):272. doi: 10.1038/s41698-025-01020-6. PMID 40764401
- [Derived] Brandt A, Klinghammer K, Schultheiss C, Paschold L, Wickenhauser C, Bauer M, Bergqvist A, Hahn D, Schafhausen P, Tometten M, Blaurock M, Zech HB, Busch CJ, Dietz A, Muller-Richter U, Alt J, Boehm A, Kowoll S, Steighardt J, Lasch A, Westgaard IH, Westhrin M, Stein A, Hinke A, Binder M. UV1 vaccination in pembrolizumab-treated patients with recurrent or metastatic head and neck cancer: A randomized multicenter phase 2 trial. Med. 2025 Jul 11;6(7):100647. doi: 10.1016/j.medj.2025.100647. Epub 2025 Apr 11. PMID 40220758
- [Derived] Brandt A, Schultheiss C, Klinghammer K, Schafhausen P, Busch CJ, Blaurock M, Hinke A, Tometten M, Dietz A, Muller-Richter U, Hahn D, Alt J, Stein A, Binder M. Tolerability and efficacy of the cancer vaccine UV1 in patients with recurrent or metastatic PD-L1 positive head and neck squamous cell carcinoma planned for first-line treatment with pembrolizumab - the randomized phase 2 FOCUS trial. Front Oncol. 2024 Feb 7;14:1283266. doi: 10.3389/fonc.2024.1283266. eCollection 2024. PMID 38384801